CLINICAL TRIAL: NCT00969111
Title: Postoperative or Salvage Radiotherapy for Node Negative Prostate Cancer Following Radical Prostatectomy
Brief Title: Postoperative or Salvage Radiotherapy (RT) for Node Negative Prostate Cancer Following Radical Prostatectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Proton Collaborative Group (Network)
Collaborators: University of Florida Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GU010-18; UFPTI 0902-PR06 (Other: University of Florida Health Proton Therapy Institute)
Record Dates: First submitted 2009-08-28; First posted 2009-08-31 (Estimated); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
Keywords: Proton Radiation, Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Protons

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Postop Non-High Risk (Experimental): Proton to 66.6 CGE
  Interventions: Radiation: Proton to 66.6 CGE
- Postop High Risk (Experimental): IMRT to 45 Gy; prostate bed proton boost of 21.6 CGE
  Interventions: Radiation: IMRT to 45 Gy; prostate bed proton boost of 21.6 CGE
- Salvage Non-High Risk (Experimental): Proton to 70.2 CGE
  Interventions: Radiation: Proton (prostate bed) to 70.2 CGE
- Salvage High Risk (Experimental): IMRT to 45 Gy; proton boost to prostate bed to 25.2 CGE
  Interventions: Radiation: IMRT to 45 Gy; proton boost to prostate bed to 25.2 CGE

INTERVENTIONS:
Radiation: IMRT to 45 Gy; prostate bed proton boost of 21.6 CGE — Postop High Risk
  Arms: Postop High Risk
Radiation: Proton (prostate bed) to 70.2 CGE — Salvage Non-High Risk
  Arms: Salvage Non-High Risk
Radiation: IMRT to 45 Gy; proton boost to prostate bed to 25.2 CGE — Salvage High Risk
  Arms: Salvage High Risk
Radiation: Proton to 66.6 CGE — Post-Op Non High Risk
  Arms: Postop Non-High Risk

SUMMARY:
The purpose of this study is to see what effects, good and/or bad, proton radiation, and/or conventional radiation and hormonal therapy (if applicable), has on prostate cancer that has already returned or the risk of prostate cancer returning.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer treated primarily with open, laparoscopic or robotically assisted prostatectomy.
* Maximum PSA value of 20 ng/ml.

Exclusion Criteria:

* Evidence of distant metastasis (M1).
* Prior systemic chemotherapy for any reason.
* Previous irradiation to the pelvis that would compromise the ability to deliver the prescribed study treatment.
* Active inflammatory bowel disease (Crohn's disease, diverticulitis or ulcerative colitis) affecting the rectum. (Non-active diverticulitis and Crohn's disease not affecting the rectum are allowed).
* History of hip replacement.
* Prior or concurrent cancer, other than non-melanomatous skin cancer, unless disease free for at least 5 years.
* Taking Saw Palmetto or methotrexate and unable or unwilling to discontinue its use during radiation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2009-08; Primary Completion 2031-08 (Estimated); Study Completion 2050-08 (Estimated)

PRIMARY OUTCOMES:
The treatment-related rate of acute grade 3 gastrointestinal and genitourinary toxicity following treatment with proton based radiation therapy. | 6 months after the end of radiation therapy

SECONDARY OUTCOMES:
Collect and analyze quality of life, treatment-related morbidity, disease control and survival outcome parameters | After radiation: every 6 months for 3 years, then annually for 20 years

CONTACTS AND LOCATIONS:
Overall Officials: Randal H Henderson, MD, Principal Investigator — University of Florida Proton Therapy Institute
Locations (4):
- United States (4):
  - Proton Center of Arkansas, Little Rock, Arkansas
  - University of Florida Proton Therapy Institute, Jacksonville, Florida
  - Northwestern Medicine Chicago Proton Center, Warrenville, Illinois
  - Inova Schar Cancer Institute, Fairfax, Virginia

REFERENCES:
- [Background] American Cancer Society. 2007. Ref Type: Electronic Citation
- [Background] Thompson IM Jr, Tangen CM, Paradelo J, Lucia MS, Miller G, Troyer D, Messing E, Forman J, Chin J, Swanson G, Canby-Hagino E, Crawford ED. Adjuvant radiotherapy for pathologically advanced prostate cancer: a randomized clinical trial. JAMA. 2006 Nov 15;296(19):2329-35. doi: 10.1001/jama.296.19.2329. PMID 17105795
- [Background] Bott SR, Freeman AA, Stenning S, Cohen J, Parkinson MC. Radical prostatectomy: pathology findings in 1001 cases compared with other major series and over time. BJU Int. 2005 Jan;95(1):34-9. doi: 10.1111/j.1464-410X.2005.05245.x. PMID 15638892
- [Background] Thompson IM, Tangen CM, Paradelo J, Lucia MS, Miller G, Troyer D, Messing E, Forman J, Chin J, Swanson G, Canby-Hagino E, Crawford ED. Adjuvant radiotherapy for pathological T3N0M0 prostate cancer significantly reduces risk of metastases and improves survival: long-term followup of a randomized clinical trial. J Urol. 2009 Mar;181(3):956-62. doi: 10.1016/j.juro.2008.11.032. Epub 2009 Jan 23. PMID 19167731
- [Background] Bolla M, van Poppel H, Collette L, van Cangh P, Vekemans K, Da Pozzo L, de Reijke TM, Verbaeys A, Bosset JF, van Velthoven R, Marechal JM, Scalliet P, Haustermans K, Pierart M; European Organization for Research and Treatment of Cancer. Postoperative radiotherapy after radical prostatectomy: a randomised controlled trial (EORTC trial 22911). Lancet. 2005 Aug 13-19;366(9485):572-8. doi: 10.1016/S0140-6736(05)67101-2. PMID 16099293
- [Background] Bianco FJ Jr, Scardino PT, Eastham JA. Radical prostatectomy: long-term cancer control and recovery of sexual and urinary function ("trifecta"). Urology. 2005 Nov;66(5 Suppl):83-94. doi: 10.1016/j.urology.2005.06.116. PMID 16194712
- [Background] Stephenson AJ, Scardino PT, Kattan MW, Pisansky TM, Slawin KM, Klein EA, Anscher MS, Michalski JM, Sandler HM, Lin DW, Forman JD, Zelefsky MJ, Kestin LL, Roehrborn CG, Catton CN, DeWeese TL, Liauw SL, Valicenti RK, Kuban DA, Pollack A. Predicting the outcome of salvage radiation therapy for recurrent prostate cancer after radical prostatectomy. J Clin Oncol. 2007 May 20;25(15):2035-41. doi: 10.1200/JCO.2006.08.9607. PMID 17513807
- [Background] Dearnaley DP, Hall E, Lawrence D, Huddart RA, Eeles R, Nutting CM, Gadd J, Warrington A, Bidmead M, Horwich A. Phase III pilot study of dose escalation using conformal radiotherapy in prostate cancer: PSA control and side effects. Br J Cancer. 2005 Feb 14;92(3):488-98. doi: 10.1038/sj.bjc.6602301. PMID 15685244
- [Background] Pollack A, Zagars GK, Starkschall G, Antolak JA, Lee JJ, Huang E, von Eschenbach AC, Kuban DA, Rosen I. Prostate cancer radiation dose response: results of the M. D. Anderson phase III randomized trial. Int J Radiat Oncol Biol Phys. 2002 Aug 1;53(5):1097-105. doi: 10.1016/s0360-3016(02)02829-8. PMID 12128107
- [Background] Sathya JR, Davis IR, Julian JA, Guo Q, Daya D, Dayes IS, Lukka HR, Levine M. Randomized trial comparing iridium implant plus external-beam radiation therapy with external-beam radiation therapy alone in node-negative locally advanced cancer of the prostate. J Clin Oncol. 2005 Feb 20;23(6):1192-9. doi: 10.1200/JCO.2005.06.154. PMID 15718316
- [Background] Shipley WU, Verhey LJ, Munzenrider JE, Suit HD, Urie MM, McManus PL, Young RH, Shipley JW, Zietman AL, Biggs PJ, et al. Advanced prostate cancer: the results of a randomized comparative trial of high dose irradiation boosting with conformal protons compared with conventional dose irradiation using photons alone. Int J Radiat Oncol Biol Phys. 1995 Apr 30;32(1):3-12. doi: 10.1016/0360-3016(95)00063-5. PMID 7721636
- [Background] Zietman AL, DeSilvio ML, Slater JD, Rossi CJ Jr, Miller DW, Adams JA, Shipley WU. Comparison of conventional-dose vs high-dose conformal radiation therapy in clinically localized adenocarcinoma of the prostate: a randomized controlled trial. JAMA. 2005 Sep 14;294(10):1233-9. doi: 10.1001/jama.294.10.1233. PMID 16160131
- [Background] Swanson GP, Hussey MA, Tangen CM, Chin J, Messing E, Canby-Hagino E, Forman JD, Thompson IM, Crawford ED; SWOG 8794. Predominant treatment failure in postprostatectomy patients is local: analysis of patterns of treatment failure in SWOG 8794. J Clin Oncol. 2007 Jun 1;25(16):2225-9. doi: 10.1200/JCO.2006.09.6495. PMID 17538167
- [Background] King CR, Kapp DS. Radiotherapy after prostatectomy: is the evidence for dose escalation out there? Int J Radiat Oncol Biol Phys. 2008 Jun 1;71(2):346-50. doi: 10.1016/j.ijrobp.2007.10.008. Epub 2008 Jan 30. PMID 18234451
- [Background] King CR, Spiotto MT. Improved outcomes with higher doses for salvage radiotherapy after prostatectomy. Int J Radiat Oncol Biol Phys. 2008 May 1;71(1):23-7. doi: 10.1016/j.ijrobp.2007.09.047. Epub 2008 Jan 22. PMID 18207668
- [Background] Feng M, Hanlon AL, Pisansky TM, Kuban D, Catton CN, Michalski JM, Zelefsky MJ, Kupelian PA, Pollack A, Kestin LL, Valicenti RK, DeWeese TL, Sandler HM. Predictive factors for late genitourinary and gastrointestinal toxicity in patients with prostate cancer treated with adjuvant or salvage radiotherapy. Int J Radiat Oncol Biol Phys. 2007 Aug 1;68(5):1417-23. doi: 10.1016/j.ijrobp.2007.01.049. Epub 2007 Apr 6. PMID 17418972
- [Background] Vargas C, Fryer A, Mahajan C, Indelicato D, Horne D, Chellini A, McKenzie C, Lawlor P, Henderson R, Li Z, Lin L, Olivier K, Keole S. Dose-volume comparison of proton therapy and intensity-modulated radiotherapy for prostate cancer. Int J Radiat Oncol Biol Phys. 2008 Mar 1;70(3):744-51. doi: 10.1016/j.ijrobp.2007.07.2335. Epub 2007 Sep 27. PMID 17904306
- [Background] Slater JD, Rossi CJ Jr, Yonemoto LT, Bush DA, Jabola BR, Levy RP, Grove RI, Preston W, Slater JM. Proton therapy for prostate cancer: the initial Loma Linda University experience. Int J Radiat Oncol Biol Phys. 2004 Jun 1;59(2):348-52. doi: 10.1016/j.ijrobp.2003.10.011. PMID 15145147
- [Background] Partin AW, Mangold LA, Lamm DM, Walsh PC, Epstein JI, Pearson JD. Contemporary update of prostate cancer staging nomograms (Partin Tables) for the new millennium. Urology. 2001 Dec;58(6):843-8. doi: 10.1016/s0090-4295(01)01441-8. PMID 11744442
- [Background] Spiotto MT, Hancock SL, King CR. Radiotherapy after prostatectomy: improved biochemical relapse-free survival with whole pelvic compared with prostate bed only for high-risk patients. Int J Radiat Oncol Biol Phys. 2007 Sep 1;69(1):54-61. doi: 10.1016/j.ijrobp.2007.02.035. Epub 2007 Apr 24. PMID 17459606
- [Background] Bolla M, Collette L, Blank L, Warde P, Dubois JB, Mirimanoff RO, Storme G, Bernier J, Kuten A, Sternberg C, Mattelaer J, Lopez Torecilla J, Pfeffer JR, Lino Cutajar C, Zurlo A, Pierart M. Long-term results with immediate androgen suppression and external irradiation in patients with locally advanced prostate cancer (an EORTC study): a phase III randomised trial. Lancet. 2002 Jul 13;360(9327):103-6. doi: 10.1016/s0140-6736(02)09408-4. PMID 12126818
- [Background] Crook J, Ludgate C, Malone S, Lim J, Perry G, Eapen L, Bowen J, Robertson S, Lockwood G. Report of a multicenter Canadian phase III randomized trial of 3 months vs. 8 months neoadjuvant androgen deprivation before standard-dose radiotherapy for clinically localized prostate cancer. Int J Radiat Oncol Biol Phys. 2004 Sep 1;60(1):15-23. doi: 10.1016/j.ijrobp.2004.02.022. PMID 15337535
- [Background] D'Amico AV, Manola J, Loffredo M, Renshaw AA, DellaCroce A, Kantoff PW. 6-month androgen suppression plus radiation therapy vs radiation therapy alone for patients with clinically localized prostate cancer: a randomized controlled trial. JAMA. 2004 Aug 18;292(7):821-7. doi: 10.1001/jama.292.7.821. PMID 15315996
- [Background] Hanks GE, Pajak TF, Porter A, Grignon D, Brereton H, Venkatesan V, Horwitz EM, Lawton C, Rosenthal SA, Sandler HM, Shipley WU; Radiation Therapy Oncology Group. Phase III trial of long-term adjuvant androgen deprivation after neoadjuvant hormonal cytoreduction and radiotherapy in locally advanced carcinoma of the prostate: the Radiation Therapy Oncology Group Protocol 92-02. J Clin Oncol. 2003 Nov 1;21(21):3972-8. doi: 10.1200/JCO.2003.11.023. PMID 14581419
- [Background] Pilepich MV, Winter K, John MJ, Mesic JB, Sause W, Rubin P, Lawton C, Machtay M, Grignon D. Phase III radiation therapy oncology group (RTOG) trial 86-10 of androgen deprivation adjuvant to definitive radiotherapy in locally advanced carcinoma of the prostate. Int J Radiat Oncol Biol Phys. 2001 Aug 1;50(5):1243-52. doi: 10.1016/s0360-3016(01)01579-6. PMID 11483335
- [Background] Pilepich MV, Winter K, Lawton CA, Krisch RE, Wolkov HB, Movsas B, Hug EB, Asbell SO, Grignon D. Androgen suppression adjuvant to definitive radiotherapy in prostate carcinoma--long-term results of phase III RTOG 85-31. Int J Radiat Oncol Biol Phys. 2005 Apr 1;61(5):1285-90. doi: 10.1016/j.ijrobp.2004.08.047. PMID 15817329
- [Background] Roach M 3rd, DeSilvio M, Lawton C, Uhl V, Machtay M, Seider MJ, Rotman M, Jones C, Asbell SO, Valicenti RK, Han S, Thomas CR Jr, Shipley WS; Radiation Therapy Oncology Group 9413. Phase III trial comparing whole-pelvic versus prostate-only radiotherapy and neoadjuvant versus adjuvant combined androgen suppression: Radiation Therapy Oncology Group 9413. J Clin Oncol. 2003 May 15;21(10):1904-11. doi: 10.1200/JCO.2003.05.004. PMID 12743142
- [Background] Denham JW, Steigler A, Lamb DS, Joseph D, Mameghan H, Turner S, Matthews J, Franklin I, Atkinson C, North J, Poulsen M, Christie D, Spry NA, Tai KH, Wynne C, Duchesne G, Kovacev O, D'Este C; Trans-Tasman Radiation Oncology Group. Short-term androgen deprivation and radiotherapy for locally advanced prostate cancer: results from the Trans-Tasman Radiation Oncology Group 96.01 randomised controlled trial. Lancet Oncol. 2005 Nov;6(11):841-50. doi: 10.1016/S1470-2045(05)70348-X. PMID 16257791
- [Background] Ghilezan MJ, Jaffray DA, Siewerdsen JH, Van Herk M, Shetty A, Sharpe MB, Zafar Jafri S, Vicini FA, Matter RC, Brabbins DS, Martinez AA. Prostate gland motion assessed with cine-magnetic resonance imaging (cine-MRI). Int J Radiat Oncol Biol Phys. 2005 Jun 1;62(2):406-17. doi: 10.1016/j.ijrobp.2003.10.017. PMID 15890582
- [Background] Padhani AR, Khoo VS, Suckling J, Husband JE, Leach MO, Dearnaley DP. Evaluating the effect of rectal distension and rectal movement on prostate gland position using cine MRI. Int J Radiat Oncol Biol Phys. 1999 Jun 1;44(3):525-33. doi: 10.1016/s0360-3016(99)00040-1. PMID 10348281
- [Background] Litzenberg D, Dawson LA, Sandler H, Sanda MG, McShan DL, Ten Haken RK, Lam KL, Brock KK, Balter JM. Daily prostate targeting using implanted radiopaque markers. Int J Radiat Oncol Biol Phys. 2002 Mar 1;52(3):699-703. doi: 10.1016/s0360-3016(01)02654-2. PMID 11849792
- [Background] Litzenberg DW, Balter JM, Hadley SW, Sandler HM, Willoughby TR, Kupelian PA, Levine L. Influence of intrafraction motion on margins for prostate radiotherapy. Int J Radiat Oncol Biol Phys. 2006 Jun 1;65(2):548-53. doi: 10.1016/j.ijrobp.2005.12.033. Epub 2006 Mar 20. PMID 16545919
- [Background] Vargas C, Yan D, Kestin LL, Krauss D, Lockman DM, Brabbins DS, Martinez AA. Phase II dose escalation study of image-guided adaptive radiotherapy for prostate cancer: use of dose-volume constraints to achieve rectal isotoxicity. Int J Radiat Oncol Biol Phys. 2005 Sep 1;63(1):141-9. doi: 10.1016/j.ijrobp.2004.12.017. PMID 16111582
- [Background] Vargas C, Martinez A, Kestin LL, Yan D, Grills I, Brabbins DS, Lockman DM, Liang J, Gustafson GS, Chen PY, Vicini FA, Wong JW. Dose-volume analysis of predictors for chronic rectal toxicity after treatment of prostate cancer with adaptive image-guided radiotherapy. Int J Radiat Oncol Biol Phys. 2005 Aug 1;62(5):1297-308. doi: 10.1016/j.ijrobp.2004.12.052. PMID 16029785
- [Background] Taylor A, Rockall AG, Reznek RH, Powell ME. Mapping pelvic lymph nodes: guidelines for delineation in intensity-modulated radiotherapy. Int J Radiat Oncol Biol Phys. 2005 Dec 1;63(5):1604-12. doi: 10.1016/j.ijrobp.2005.05.062. Epub 2005 Sep 29. PMID 16198509
- [Background] Ehrenpreis ED, Jani A, Levitsky J, Ahn J, Hong J. A prospective, randomized, double-blind, placebo-controlled trial of retinol palmitate (vitamin A) for symptomatic chronic radiation proctopathy. Dis Colon Rectum. 2005 Jan;48(1):1-8. doi: 10.1007/s10350-004-0821-7. PMID 15690650
- [Background] Denton A, Forbes A, Andreyev J, Maher EJ. Non surgical interventions for late radiation proctitis in patients who have received radical radiotherapy to the pelvis. Cochrane Database Syst Rev. 2002;(1):CD003455. doi: 10.1002/14651858.CD003455. PMID 11869662
- [Background] Cavcic J, Turcic J, Martinac P, Jelincic Z, Zupancic B, Panijan-Pezerovic R, Unusic J. Metronidazole in the treatment of chronic radiation proctitis: clinical trial. Croat Med J. 2000 Sep;41(3):314-8. PMID 10962052
- [Background] Delanian S, Lefaix JL. Current management for late normal tissue injury: radiation-induced fibrosis and necrosis. Semin Radiat Oncol. 2007 Apr;17(2):99-107. doi: 10.1016/j.semradonc.2006.11.006. PMID 17395040
- [Background] Lefaix JL, Delanian S, Vozenin MC, Leplat JJ, Tricaud Y, Martin M. Striking regression of subcutaneous fibrosis induced by high doses of gamma rays using a combination of pentoxifylline and alpha-tocopherol: an experimental study. Int J Radiat Oncol Biol Phys. 1999 Mar 1;43(4):839-47. doi: 10.1016/s0360-3016(98)00419-2. PMID 10098440
- [Background] Delanian S, Porcher R, Balla-Mekias S, Lefaix JL. Randomized, placebo-controlled trial of combined pentoxifylline and tocopherol for regression of superficial radiation-induced fibrosis. J Clin Oncol. 2003 Jul 1;21(13):2545-50. doi: 10.1200/JCO.2003.06.064. PMID 12829674
- [Background] Spry N, Halkett G, Aoun S, Spry J, Yeoh E. Development of a European organization for research and treatment of cancer module to assess the quality of life of patients with proctitis after pelvic radiotherapy for malignancy. Int J Radiat Oncol Biol Phys. 2008 Oct 1;72(2):522-8. doi: 10.1016/j.ijrobp.2007.12.062. Epub 2008 Apr 18. PMID 18374505